CLINICAL TRIAL: NCT03921047
Title: Characterization of T-cell Repertoire in Patients With AML Undergoing HSCT Through Next-Generation Sequencing of T Cell Receptor Alpha (TCRA) and T Cell Receptor Beta (TCRB) Genes
Brief Title: Characterization of T-cell Repertoire in Patients With Acute Myeloid Leukemia Undergoing Donor Stem Cell Transplant
Status: Recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 9L-16-10; NCI-2017-02440 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9L-16-10 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ancillary-correlative (next generation sequencing): Patents undergo collection of blood samples before, on day 100, and 1 year after HSCT. Donors undergo collection of blood at the time of HSCT for RNA-based next generation sequencing of TCRA and TCRB genes.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research trial studies characterization of T-cell repertoire through next-generation sequencing in patients with acute myeloid leukemia undergoing stem cell transplant. Characterizing T-cell repertoire may help to understand if immune system plays a significant role in high risk patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Characterize the T cell receptor (TCR) repertoire in acute myeloid leukemia (AML) patients before and after receiving hematologic stem cell transplantation (HSCT).

II. Identify molecular changes (germline variants and somatic mutations) that contribute to shaping the TCR repertoire.

OUTLINE:

Patents undergo collection of blood samples before, on day 100, and 1 year after HSCT. Donors undergo collection of blood at the time of HSCT for ribonucleic acid (RNA)-based next generation sequencing of TCRA and TCRB genes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML scheduled to undergo HSCT at University of Southern California (USC)

Exclusion Criteria:

* Inability to provide consent because of severe mental disorders
* Donor unwilling to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AML scheduled to undergo HSCT
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-04-12 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Time to diagnosis of acute graft versus (vs.) host disease (aGVHD) | Up to 4 years
  Will be calculated as the time from stem cell infusion until the date of the diagnosis of aGVHD. If a patient dies prior to day 100 and does not have aGVHD, the patient will be censored at the time of death; all patients without aGVHD will be censored on day 100.
Time to diagnosis of relapse | Up to 4 years
  Will be calculated as the time from stem cell infusion until the date of the of the diagnosis of relapse Patients who die of treatment toxicity or other cause, prior to relapse, will be censored at the time of death; all patients will be censored at 365 days following transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Houda Alachkar, PharmD, PhD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States